CLINICAL TRIAL: NCT02479750
Title: Evaluation of ColdZyme® on Experimentally Induced Common Cold. -A Double-blind, Randomized, Placebo-controlled Study in Healthy Volunteers.
Brief Title: Evaluation of ColdZyme® on Experimentally Induced Common Cold.
Acronym: COLDPREVII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Enzymatica AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENZY-002
Record Dates: First submitted 2015-06-22; First posted 2015-06-24 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ColdZyme (Experimental): ColdZyme® mouth spray liquid. Treatment (6 doses per day) will be applied for 11 days from the day of inoculation.
  Interventions: Device: ColdZyme® mouth spray
- Placebo (Placebo Comparator): Sugar based mouth spray liquid manufactured to mimic ColdZyme® mouth spray. Treatment (6 doses per day) will be applied for 11 days from the day of inoculation.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: ColdZyme® mouth spray
  Arms: ColdZyme
Device: Placebo
  Arms: Placebo

SUMMARY:
This study evaluates the performance of ColdZyme® mouth spray on prevention of common cold symptoms on experimentally induced rhinovirus upper respiratory tract infection in healthy volunteers. Half of participants will receive ColdZyme® mouth spray while the other half will receive placebo.

DETAILED DESCRIPTION:
88 subjects will be inoculated with rhinovirus 16 via the nasal route. The subjects will be randomized 1:1 to ColdZyme® or placebo. Treatment (6 doses per day) will be applied for 11 days from the day of inoculation. The subjects will visit the investigational clinic on 6 occasions. During these visits the subjects will leave nasal (lavage) and pharyngeal (swab) samples for quantification of virus replication. All subjects will have a diary for scoring of cold symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects between 16-70 years. The investigator judges the definition of healthy by detailed medical history and physical examination.
* Females of childbearing potential: shall use reliable method of birth control. Reliable methods are hormonal contraceptives (combination pills, injections or implants), intrauterine device, condom or declared absence of sexual contact. Post-menopausal woman is defined as absence of menstrual discharge for at least two years.
* Signed informed consent form prior to any study-related procedures.
* Willingness and ability to adhere to the prohibitions and restrictions specified in this protocol.
* Perceived to have had at least one cold per year

Exclusion Criteria:

* Smoker, during the last 12 months
* Any cold symptom within the last month such as sore throat, sneezing, rhinorrhoea, malaise, nasal obstruction or cough.
* Presence (at screening) of serum rhinovirus 16 neutralising antibody titers at greater than or equal to one in two dilution.
* Active allergic rhinitis, asthma or chronic obstructive pulmonary disease during study period.
* Nasal disease, e.g. nasal polyposis, significant septal deviation, chronic rhinosinusitis, etc.
* Females: Pregnant, breast-feeding or intentions to become pregnant during the study.
* Evidence or history of drug or alcohol abuse.
* Use of any prescribed or non-prescribed medication (except for contraceptives, paracetamol and ibuprofen) within 2 weeks prior to the first administration of investigational product.
* Use of any over the counter cold prophylaxis products such as ColdZyme®, C-vitamins, zinc or Echinacea within 1 month prior to the first administration of investigational product.
* Participation in other clinical trial with medical investigational product within 60 days prior to the first administration of investigational product.
* Hypersensitivity/allergy to any of the device ingredients
* Individuals with close contact to at risk patient group:
* infants (less than 6 months);
* the extremely elderly or infirm;
* pregnant women;
* patients with severe lung disease (asthma/cystic fibrosis (CF)/COPD);
* patients with immunosuppression.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2016-07-25 (Actual); Study Completion 2016-07-25 (Actual)

PRIMARY OUTCOMES:
Reduction of virus load | 7 days
  The primary objective is to investigate the protective effect of ColdZyme® mouth spray against infection in the oropharynx by common cold virus (rhinovirus 16) in vivo in relation to placebo

SECONDARY OUTCOMES:
Reduce the number of days with common cold symptoms | 11 days
Reduce the number of days with virus present in oropharynx | 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Mallia, MD, Principal Investigator — NHLI, Imperial College
Locations (1):
- National Heart and Lung Institute, Imperial College, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No